CLINICAL TRIAL: NCT03125993
Title: Effects of Brisk Walking on Overweight/Obesity Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Center for Disease Prevention and Control (Other Government)
Responsible Party: Principal Investigator, Xue-yan Zheng, Dr., Guangdong Center for Disease Prevention and Control
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BWOE
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: obesity; brisk walking
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This study is a prospective 4-month follow-up scheme in which patients were treated with the following intervention: > 10000 steps, > five days, per week. For individual follow-up, body components and metabolic risk factors will be tested before and after the study. Every participants will be followed up in community visits every month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- >10000 steps brisk walking (Experimental): This study is a prospective 4-month follow-up scheme in which patients were treated with the following intervention: > 10000 steps, > five days, per week. For individual follow-up, body components and metabolic risk factors will be tested before and after the study.
  Interventions: Behavioral: >10000 steps brisk walking

INTERVENTIONS:
Behavioral: >10000 steps brisk walking — This study is a prospective 4-month follow-up scheme in which patients were treated with the following intervention: > 10000 steps, > five days, per week brisk walking.

SUMMARY:
1.Objective

The investigators aim to determine the effect of brisk walking prescription (> 10000 steps, > five days, per week) on body components and metabolic risk factors among patients with overweight/obesity. The objectives are as follow:

1. The body components changes before/after the brisk walking prescription (> 10000 steps, > five days per week) intervention in overweight/obesity population;
2. The metabolic risk factors changes before/after the brisk walking prescription (<10000 steps or <five days per week) intervention in overweight/obesity population

2.Study design This study is a prospective 4-month follow-up scheme in which patients were treated with the following intervention: > 10000 steps, > five days, per week. For individual follow-up, body components and metabolic risk factors will be tested before and after the study. Every participants will be followed up in community visits every month.

3. Statistical analysis Statistical analysis will be performed using SPSS 16.0 version package (SPSS Inc., Chicago, IL.). Numerical data will be presented as mean ± standard deviation for normal distribution or otherwise median (interquartile range). Two-sided independent t-test is adopted for between-group comparison on end-points with normal distribution, otherwise non-parametric test. Row-Column table will be analyzed through chi-square test. P<0.05 is taken as statistical significant.

DETAILED DESCRIPTION:
Obesity/overweight has been recognized as one of the most important global health threats worldwide, which is closely related to metabolism syndrome including insulin resistance, hypertension, dyslipidemia and hyperglycemia.

In 2013, an estimated 36.9% of men and 38.0% of women were overweight (BMI >25 kg/m2) worldwide, with attributable fractions for CHD as high as 25% in the United States and 58% in the Asia-Pacific Region. Furthermore, a strong and continuous association between body mass index (BMI) and coronary heart disease (CHD) has been reported for values of BMI above 20kg/m2 .

Numerous studies have recognized the role of physical activity in promoting moderate weight loss, weight loss maintenance, and having broad-reaching implications for cardiovascular disease mortality indices, as well as reducing healthcare expenditures. The findings of a recent review suggest that mild-to-moderate intensity exercises that include both aerobic and resistance training result in additional metabolic benefits in people with obesity or type 2 diabetes. Although weight loss is minimal, body composition improves. Brisk walking, at an individual level, prove to be the physical activity most easy to maintain and could be progressively increased in intensity, achieving a cardiorespiratory benefit and decrease adiposity in the unfit.

Several small clinical trials reported inconsistent findings of short-term exercise programs on brisk walking among patients with overweight/obesity. However, these studies did not provide comparable indices, duration and intensity. Furthermore, the brisk walking effect of current physical activity guidelines on obesity/overweight is uncertain.

The current study aimed to evaluate the effects of brisk walking ( > 10000 steps, > five days, per week) on body components and metabolic risk factors among patients with overweight/obesity.

ELIGIBILITY:
Inclusion Criteria:

1. The inclusion criterion is individual with sedentary behaviors, adding any of the following behavior:

   1. individuals with BMI ≥24 kg/m2
   2. waist circumstance ≥102cm in male; waist circumstance ≥88cm in female;
   3. waist circumstance/hip circumstance>1.0 in male; waist circumstance/hip circumstance> 0.9 in female.

Exclusion Criteria:

- Participants were excluded with the presence of significant cardiac or pulmonary disease that could result in hypoxia or decreased perfusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-04-25 (Estimated); Primary Completion 2017-08-25 (Estimated); Study Completion 2017-08-30 (Estimated)

PRIMARY OUTCOMES:
BMI | Change from Baseline BMI at 4 months
  Body components

SECONDARY OUTCOMES:
Systolic blood pressure | Change from systolic blood pressure at 4 months
  Cardiovascular risk factors
Diastolic blood pressure | Change from diastolic blood pressure at 4 months
  Cardiovascular risk factors
Plasma glucose | Change from Plasma glucose at 4 months
  Cardiovascular risk factors
visceral fat | Change from visceral fat at 4 months
  Cardiovascular risk factors
serum triglycerides | Change from serum triglycerides at 4 months
  Cardiovascular risk factors
serum total cholesterol | Change from serum total cholesterol at 4 months
  Cardiovascular risk factors
high density lipoprotein-C | Change from high density lipoprotein-C at 4 months
  Cardiovascular risk factors
low density lipoprotein-C | Change from low density lipoprotein-C at 4 months
  Cardiovascular risk factors
heart rate | Change from heart rate at 4 months
  Cardiovascular risk factors
abdominal circumstance | Change from abdominal circumstance at 4 months
  Body components
body fat percentage | Change from body fat percentage at 4 months
  Body components
visceral fat percentage | Change from visceral fat percentage at 4 months
  Body components
waist circumstance/hip circumstance | Change from waist circumstance/hip circumstance at 4 months
  Body components

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared with other researchers, for data safety.

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] Hubert HB, Feinleib M, McNamara PM, Castelli WP. Obesity as an independent risk factor for cardiovascular disease: a 26-year follow-up of participants in the Framingham Heart Study. Circulation. 1983 May;67(5):968-77. doi: 10.1161/01.cir.67.5.968. PMID 6219830
- [Background] Lee CM, Colagiuri S, Ezzati M, Woodward M. The burden of cardiovascular disease associated with high body mass index in the Asia-Pacific region. Obes Rev. 2011 May;12(5):e454-9. doi: 10.1111/j.1467-789X.2010.00849.x. Epub 2011 Mar 2. PMID 21366838
- [Background] Swift DL, Johannsen NM, Lavie CJ, Earnest CP, Church TS. The role of exercise and physical activity in weight loss and maintenance. Prog Cardiovasc Dis. 2014 Jan-Feb;56(4):441-7. doi: 10.1016/j.pcad.2013.09.012. Epub 2013 Oct 11. PMID 24438736
- [Background] Hills AP, Shultz SP, Soares MJ, Byrne NM, Hunter GR, King NA, Misra A. Resistance training for obese, type 2 diabetic adults: a review of the evidence. Obes Rev. 2010 Oct;11(10):740-9. doi: 10.1111/j.1467-789X.2009.00692.x. PMID 20003071
- [Background] Hills AP, Byrne NM, Wearing S, Armstrong T. Validation of the intensity of walking for pleasure in obese adults. Prev Med. 2006 Jan;42(1):47-50. doi: 10.1016/j.ypmed.2005.10.010. Epub 2005 Dec 1. PMID 16325248
- [Background] Williams PT. Association between walking distance and percentiles of body mass index in older and younger men. Br J Sports Med. 2008 May;42(5):352-6. doi: 10.1136/bjsm.2007.041822. Epub 2008 Apr 2. PMID 18385193
- [Background] Ikenaga M, Yamada Y, Kose Y, Morimura K, Higaki Y, Kiyonaga A, Tanaka H; Nakagawa Study Group. Effects of a 12-week, short-interval, intermittent, low-intensity, slow-jogging program on skeletal muscle, fat infiltration, and fitness in older adults: randomized controlled trial. Eur J Appl Physiol. 2017 Jan;117(1):7-15. doi: 10.1007/s00421-016-3493-9. Epub 2016 Nov 15. PMID 27848017
- [Background] Schutz Y, Nguyen DM, Byrne NM, Hills AP. Effectiveness of three different walking prescription durations on total physical activity in normal- and overweight women. Obes Facts. 2014;7(4):264-73. doi: 10.1159/000365833. Epub 2014 Aug 1. PMID 25137221
- [Background] Takahashi PY, Quigg SM, Croghan IT, Schroeder DR, Ebbert JO. Effect of pedometer use and goal setting on walking and functional status in overweight adults with multimorbidity: a crossover clinical trial. Clin Interv Aging. 2016 Sep 1;11:1099-106. doi: 10.2147/CIA.S107626. eCollection 2016. PMID 27621602